CLINICAL TRIAL: NCT04028076
Title: Peers LEAD: Partnering With Peers in the Community to Improve Diabetes Medication Adherence for African Americans in Madison and Milwaukee: A Pre-Post Single Group Intervention
Brief Title: Improving Diabetes Medication Adherence for African Americans in Madison and Milwaukee Through Peer Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0721; A561000 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison); Protocol Version 6/7/2020 (Other: UW Madison)
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Type2 Diabetes; Medication Adherence; Medication Nonadherence; Peer Support
Keywords: Peer Support; Type2 Diabetes; African American
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peers LEAD (Experimental): 8-week educational behavioral intervention
  Interventions: Behavioral: Peers Supporting Health-Literacy, Self Efficacy, Advocacy and Adherence

INTERVENTIONS:
Behavioral: Peers Supporting Health-Literacy, Self Efficacy, Advocacy and Adherence — An 8-week culturally appropriate educational behavioral intervention that consists of structured group diabetes education and follow-up peer support with PAs. There will be 3 separate group education sessions led by a physician, AA pharmacist and AA diabetes educator. All PAs will attend each group session to learn together with their PBs and build social interactions. Weeks 1 and 2 consist of 2-hour group education between the participants and diabetes educator, and participants and pharmacist, respectively. Pre-test intervention data including A1c will be collected in Week 1. In Weeks 3-7, PAs will deliver the intervention content to PBs over the phone as well as help them set a goal towards getting healthy. An existing video/text messaging app, called WhatsApp® will be offered as an option to use to further enhance PA-PB interaction.
  Other Names: Peers LEAD

SUMMARY:
The burden of diabetes is higher among African Americans (AAs) in Wisconsin as hospitalization rates for diabetes complications such as stroke and amputations are four times higher than whites and has worsened by 334% since 2011. The most important self-management behavior for improving diabetes outcomes is medication adherence, i.e., taking medicines as recommended by providers. Poor adherence to diabetes medications is common among AAs and contributes to disproportionally worse outcomes. While the reasons for nonadherence are multifactorial, health beliefs, lack of self-efficacy, social support, and limited health literacy, are critical factors for AAs. Due to discrimination experiences and provider distrust, AAs may have health beliefs that do not align with biomedicine. Existing adherence interventions designed for general populations may be ineffective for AAs because they do not adequately address these fundamental factors.

The intervention is peer-led, such that AAs who have diabetes and are adherent to their medicines (Peer Ambassadors- (PAs)) are paired with AAs who have diabetes and are nonadherent (Peer Buddies- PBs)).Throughout the 8-week program, PAs actively support and teach PBs about self-advocacy in patient-provider relationships, as well as sharing their experiences managing diabetes, providing social support, enhancing health literacy, patient activation (engagement and empowerment) and self-efficacy. PAs help deliver the intervention via initial face-to-face and phone/app follow-ups with PBs, in addition to structured group education delivered to PBs by a physician, pharmacist, and diabetes educator separately. The investigator's aim is to use a community-engaged design to pilot the intervention, assessing the feasibility of gathering pre/post outcomes including culturally-informed diabetes-health beliefs, self-efficacy, patient activation, medication adherence (using surveys), and A1c, and further refine the intervention via feedback from an advisory board comprised of the PAs.

The investigators hypothesize that the intervention will be feasible for AAs with diabetes. This study uses a collaborative approach involving patient stakeholders throughout the research process by directly engaging AAs with diabetes to utilize their experience, knowledge and advice. This project advances the development of culturally-appropriate medication adherence interventions for AAs with diabetes.

DETAILED DESCRIPTION:
In the United States, diabetes affects 3.7 million African Americans (AAs) who are more likely to be diagnosed compared to non-Hispanic whites and are at a greater risk for diabetes-related death and disability. Diabetes is the seventh leading cause of death in Wisconsin, incurring an estimated $3.9 billion annually in health care and lost productivity costs. Each year, more than 1,300 people in Wisconsin die from diabetes and many more suffer diabetes-related complications such as heart disease and amputations. This burden is higher among African Americans (AAs) whose hospitalization rates for diabetes-related complications are four times higher than whites. The most important self-management behavior for improving diabetes outcomes is medication adherence, i.e., taking medications according to provider recommendations. Poor medication adherence places a significant economic burden on US healthcare systems, resulting in $290 billion in costs. A nonadherent patient requires three extra medical visits per year, leading to $2000 increased treatment costs annually. In diabetes, the estimated US cost savings due to improving poor adherence is $1.16 billion. Nonadherence is thus a critical societal problem with negative economic consequences and detrimental effects on health and well-being.

Poor adherence to diabetes medicines is common among AAs and contributes to disproportionally worse diabetes outcomes for AAs. AAs have a 25% lower adherence to diabetes medications than non-Hispanic whites. While the reasons for nonadherence are multifactorial, health beliefs, lack of social support, and limited health literacy, are critical factors for AAs. Due to limited access to high quality healthcare, discrimination experiences, and distrust in providers, AAs may have health beliefs that do not align with biomedicine. Existing adherence interventions designed for general populations may be ineffective for AAs because they do not adequately address these fundamental psychosocial factors. The proposed work builds on the investigator's studies of AAs' diabetes experiences and medication adherence. The investigator's previous research showed that AAs felt a loss of autonomy because of diabetes and believed that diabetes was caused by exposure to certain medications. Navigating the healthcare system seemed difficult. Some AAs did not take their medicines because they did not know how to ask their provider questions. AAs wanted peers to support/teach self-advocacy and positive empowerment in patient-provider relationships. Hence, the investigators worked with community/patient stakeholders to develop a prototype 8-week peer-led culturally appropriate intervention to address identified psychosocial/ sociocultural issues and enhance diabetes medication adherence for AAs, called Peers Supporting Health Literacy, Self-Efficacy, Advocacy and Adherence (Peers LEAD).

Typically, peer support occurs through group, nurse and community health worker visits; however, these require expensive professional staff. Peers LEAD offers an innovative, culturally appropriate and more informal, low-cost means of providing peer support with similar benefits. The long-term goal is to decrease diabetes-related morbidity among AAs through culturally appropriate interventions to increase medication adherence. The study objective is to pilot Peers LEAD using a community-based participatory design to examine for feasibility, outcomes including culturally-informed diabetes-health beliefs, diabetes and medication self-efficacy, patient activation (a measure of engagement/empowerment), medication adherence, and blood glucose, and refine Peers LEAD via participant feedback. The central hypothesis is that Peers LEAD will be feasible and effective for AAs with diabetes, leading to improved outcomes in self-efficacy, activation, adherence, and blood glucose. The study aims are:

Aim 1: To pilot PEERS LEAD to test the feasibility and acceptability of the intervention intended to shift negative diabetes-health beliefs to positive, enhance diabetes self-efficacy, and improve adherence, and blood glucose levels. In conjunction with an interdisciplinary team of a physician, pharmacist and diabetes educator who will provide structured education, Peer Ambassador Board (PAB) members will help deliver Peers LEAD, via initial face-to-face and phone/messaging app follow-ups, serving as peer ambassadors (PAs). Peer buddies (PBs) (AAs 30-65 years old with type 2 diabetes and poor medication adherence) will participate in the program, with a target of 10 20 PBs each in Madison and 10 PBs in Milwaukee. PBs will complete surveys and glucose tests assessing changes in outcomes. Interviews and focus groups will be conducted with all PBs and PAs respectively to get feedback on the intervention. The investigators hypothesize that PA/PB feedback will lead to a feasible intervention showing improvement in adherence and glucose levels for the PBs.

Aim 2: To refine PEERS LEAD for AAs with diabetes using feedback from Peer Ambassador Boards and Peer Buddies. The investigators will: (1) establish two PABs, (2) train PAB members as PAs, (3) elicit feedback to refine Peers LEAD.

This study uses a collaborative approach involving patient stakeholders throughout the research process by directly engaging AAs with diabetes to utilize their experience, knowledge and advice. This is the first study to enhance peer support for AAs with diabetes using phone/messaging app technology. This project advances the development of innovative interventions for AAs with diabetes and focuses on social and behavioral constructs identified from the investigator's prior work to influence medication adherence.

Overall Study Design: This pilot research will be conducted in 2 phases using an intervention mixed methods design in which the investigators will test the 8-week Peers Supporting Health Literacy, Self-Efficacy, Advocacy and Adherence (Peers LEAD) intervention in Phase 1, and then examine specific intervention elements for refinement in Phase 2. The rationale for this design is that neither quantitative nor qualitative methods are sufficient in explaining the outcomes of the intervention. Mixing both methods gives a more complete analysis of Peers LEAD. Qualitative results collected during and after the intervention will allow the investigators to further explain the outcomes, examine participant's experiences and modify the methods in a follow-up and/or dissemination study.

ELIGIBILITY:
Inclusion Criteria:

Peer Ambassadors:

* Men and women 30-65 years old with type 2 diabetes who self-identify as Black/AA and can speak/read English at a 6th grade level,
* Self-report as prescribed one oral diabetes medication and are adherent to taking it (11 on the ARMS-D scale),
* Have access to/can use a phone with cellular/internet use during the study.

Peer Buddies:

* Men and women 30-65 years old with type 2 diabetes who self-identify as Black/AA and can speak/read English at a 6th grade level,
* Self-report as prescribed one oral diabetes medication and are non-adherent to taking it (greater than 11 on the ARMS-D scale)
* Have access to/can use a phone with cellular/internet use during the study.

Exclusion Criteria:

Peer Ambassadors:

* Individuals who are only using insulin (adherence may differ for these individuals)
* Individuals who report diagnosis of mental illness/psychosis.

Peer Buddies:

* Individuals who are only using insulin (adherence may differ for these individuals),
* Individuals who have a diagnosed psychiatric disorder

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | Peer Buddy's Change in Hemoglobin A1c will be measured from baseline (prior to the intervention) at 3 months
  A study team researcher with clinical experience will perform a finger prick test to collect a small amount of blood to test for hemoglobin A1C. A glucometer will be used to measure the specimen's A1c level. The research team will promptly report all A1c levels to the participant by handwriting the result on a paper.

SECONDARY OUTCOMES:
Beliefs about Medicines Questionnaire | Peer Buddies will complete a 20-minute paper survey prior to the intervention and up to 12 weeks later.
  Participant's beliefs about diabetes medicines.
Culturally adapted illness perception questionnaire | Peer Buddies will complete a 20-minute paper survey prior to the intervention and up to 12 weeks later.
  Participant's beliefs about diabetes as an illness.
Self-Efficacy for Appropriate Medication Use Scale (SEAMS) | Peer Buddies will complete a 20-minute paper survey prior to the intervention and up to 12 weeks later.
  This scale measures participant's self-efficacy related to medication use. The range of total scores is 13-39. Lower values indicate worse outcomes.
Newest Vital Sign | Peer Buddies will complete a 20-minute paper survey prior to the intervention and up to 12 weeks later.
  The Newest Vital Sign is a valid and reliable screening tool available that identifies patients at risk for low health literacy. It is a nutrition label that is accompanied by 6 questions, with total scores ranging from 0-6, with lower values indicating worse outcomes.
Adherence to Refills and Medications Scale for Diabetes (ARMS-D) | Peer Buddies will complete a 20-minute paper survey prior to the intervention and up to 12 weeks later.
  Measure of self-reported diabetes medication adherence. Total scores range from 11-44, with higher values indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka Shiyanbola, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiyanbola OO, Maurer M, Mott M, Schwerer L, Sarkarati N, Sharp LK, Ward E. A feasibility pilot trial of a peer-support educational behavioral intervention to improve diabetes medication adherence in African Americans. Pilot Feasibility Stud. 2022 Nov 14;8(1):240. doi: 10.1186/s40814-022-01198-7. PMID 36376960